CLINICAL TRIAL: NCT02547506
Title: Comparison of Cardiorespiratory Fitness Among Regular Exercisers With and Without Parkinson Disease and Across Different Modes of Group Exercise
Status: Completed | Type: Observational
Sponsor: University of Indianapolis (Other)
Responsible Party: Principal Investigator, Stephanie Miller, Professor, University of Indianapolis
Other Study IDs: 0726
Record Dates: First submitted 2015-09-09; First posted 2015-09-11 (Estimated); Last update posted 2019-10-09 (Actual); Status verified 2019-10

CONDITIONS: Parkinson Disease
Keywords: cardiorespiratory fitness; group exercise
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Parkinson Disease (Boxing): Individuals with Parkinson Disease who participate in boxing on a regular basis
- Parkinson Disease (Group Exercise): Individuals with Parkinson Disease who participate in group exercise other than boxing on a regular basis
- Healthy Controls: Individuals without disability who participate in group exercise other than boxing on a regular basis

SUMMARY:
The central goal of the proposed study is to generate essential pilot data necessary to support an established line of research leading to future extramural grant submissions. The aims of the current study are two-fold: 1) to compare cardiorespiratory fitness (CRF) and gait endurance across three groups of people: (1) individuals with Parkinson Disease (PD) who participate in boxing on a regular basis, (2) individuals with PD who participate in exercise other than boxing on a regular basis and (3) healthy controls of the same age who exercise on a regular basis and 2) to examine the relationship between CRF and motor symptoms of PD (bradykinesia, tremor and postural instability). Forty-five participants (15 for each group) who participate in exercise on a regular basis (at least 120 minutes of exercise per week for the past 3 months) will be recruited for this cross-sectional study. In a single testing session, participants will perform the following tests: (1) clinical performance measures and (2) a CRF assessment. A one-way ANOVA with appropriate post hoc tests will be used to examine differences in dependent variables across the three exercise groups. Relationships between CRF and clinical performance measures will be evaluated with Pearson's correlation coefficients.

ELIGIBILITY:
Inclusion Criteria:

* All participants included in this study must be between the ages of 55 and 75
* Be able to ambulate independently without physical assistance, assistive device, or lower extremity orthosis
* Be able to follow at least 3-step verbal commands
* Participate in a community-based group exercise program
* Be classified as regular exercisers by participating in 120 minutes per week for at least 3 months
* And have a physician's consent to undergo a graded exercise test (GXT).
* Furthermore, only participants that are identified as low or moderate risk for cardiovascular disease based on ACSM's risk stratification guidelines will be included in the study.
* Participants for the two PD groups must have a diagnosis of idiopathic PD
* Have a Hoehn-Yahr score of 1, 2, or 3
* And either participate regularly in boxing training at Rock Steady Boxing or participate in another community-based group exercise program on a regular basis, classified as 120 minutes per week for at least 3 months.

Exclusion Criteria:

* Participants may not be included in the study if they have had any surgery in the past 6 months
* Current musculoskeletal or complications from other health issues that influence walking.
* The participants without disability cannot be involved in the study if they have any preexisting neurological conditions.
* Participants with PD cannot be involved in the study if they have preexisting neurological conditions other than idiopathic PD (e.g. no diagnosis of Parkinson Plus syndrome), past brain surgery or implantation of a deep brain stimulator.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 45 individuals will be enrolled in this cross-sectional study. Three groups will each consist of 15 individuals (individuals with Parkinson Disease that participate in boxing, individuals with Parkinson disease that participate in group exercise other than boxing, and individuals without disability that participate in group exercise other than boxing).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-09; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Cardiorespiratory Fitness | 1 day
  Aerobic capacity determined via VO2max protocol

SECONDARY OUTCOMES:
Six Minute Walk Test | 1 day
  Gait endurance will be determined by having participants walk as far as they can on a pre-determined, fixed distance course of 30 meters one way, in six minutes, resting if needed.
Unified Parkinson's Disease Rating Scale | 1 day
  The MDS-UPDRS is a revision of the original UPDRS, and is a used to assess impairments related to PD. The inventory consists of multiple questions self-assessing an individual's activities of daily living (ADLs), as well as, an assessed examination of the motor symptoms associated with PD.
StepWatch Activity Monitor | 7 days
  Home and community stepping activity will be assessed using a StepWatch Activity Monitor (SAM) worn by the patient.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Indianapolis, Indianapolis, Indiana, United States